CLINICAL TRIAL: NCT05097430
Title: Enhancing HIV Pre-Exposure Prophylaxis (PrEP) by Targeting Hazardous Alcohol Use and Concurrent Conditions
Brief Title: PrEP and Alcohol - Enhancing HIV Pre-Exposure Prophylaxis (PrEP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: University Health Network, Toronto (Other); Maple Leaf Research (Other)
Responsible Party: Principal Investigator, Paul Shuper, Senior Scientist and Section Head, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 4UH3AA026212-03 (NIH)
Record Dates: First submitted 2021-09-30; First posted 2021-10-28 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Hazardous Alcohol Use
Keywords: PrEP; Alcohol; Substance use; Depression
MeSH Terms: conditions — Substance-Related Disorders; Depression | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the intervention condition or treatment as usual (TAU) based on a 2:1 intervention:TAU ratio.
Who Masked: Investigator
Masking Description: This is not a double-blind study. Participants in the intervention arm will be aware that they are receiving the intervention but the investigators will not know as the randomization will take place within the software program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alcohol-focused brief intervention (Experimental): Intervention arm participants will be provided with an electronically-delivered, personalized drinking feedback report that compares their drinking with other Canadian males of the same age. This report also includes other relevant feedback, including an assessment of severity of alcohol use, and it provides recommendations for safe levels of alcohol consumption.
  Interventions: Behavioral: Alcohol-focused brief intervention
- Treatment as usual (No Intervention): Treatment as usual (TAU) participants will not receive the intervention.

INTERVENTIONS:
Behavioral: Alcohol-focused brief intervention — The primary intervention component is the Check Your Drinking (CYD) intervention - an electronically-delivered brief intervention designed to assess and provide personalized feedback regarding the quantity, frequency, and severity of one's alcohol consumption. Additionally, intervention condition participants who are identified as having a concurrent substance use concern or who may be experiencing depression will receive information about local resources that can assist with such concerns.
  Arms: Alcohol-focused brief intervention

SUMMARY:
The present investigation entails a pilot randomized controlled trial to explore whether a stand-alone, alcohol-reduction, brief intervention (with a module on substance use and depression) would be feasible, acceptable, and potentially efficacious within the context of HIV pre-exposure prophylaxis (PrEP) treatment.

DETAILED DESCRIPTION:
Although HIV pre-exposure prophylaxis (PrEP) is an effective tool that can help prevent the acquisition of HIV, its degree of effectiveness has been shown to be linked to a number of key behaviors, including treatment adherence, attendance in follow-up care, and the concurrent use of condoms. Hazardous alcohol consumption has the potential to contribute to suboptimal PrEP adherence, poor retention in PrEP care, and condomless sex/sexually transmitted infections (STIs); and its impact on these PrEP-related behaviors may also become exacerbated in the presence of concurrent issues such as substance use and depression, thus reflecting a potential syndemic effect. The present investigation entails a pilot randomized controlled trial in which 120 hazardous drinking, PrEP-prescribed men who have sex with men (MSM) will be randomly assigned to receive either a tablet-based, alcohol-reduction brief intervention or treatment-as-usual. Participants assigned to the former condition for whom substance use- and/or depression-related concerns are identified will additionally be provided with links to relevant supportive resources. Feasibility and acceptability of the intervention will be examined. Furthermore, biomarker testing and self-report electronic surveys at baseline, 3-months, and 6-months will be employed to assess the preliminary impact of the intervention on alcohol use, PrEP adherence, retention in PrEP care, and the engagement in condomless sex/STI acquisition.

ELIGIBILITY:
Inclusion Criteria: Participants must be:

* aged 18 years or older,
* be a patient of Toronto General Hospital (TGH) or Maple Leaf Medical Clinic (MLMC),
* be a man who identifies as gay, bisexual, and/or a man who has sex with other men,
* have been prescribed PrEP for at least 3 months, and
* meet the criteria for hazardous drinking, (i.e., based on a score of ≥4 on the Alcohol Use Disorders Identification Test-Consumption measures (AUDIT-C)).

Exclusion Criteria:

* Participants will be excluded if they do not meet all of the above-mentioned inclusion criteria.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study only includes men who have sex with men. This criterion is based on the fact that in Canada and the United States, men who have sex with men (MSM) remain the risk group most affected by HIV, comprising roughly two-thirds of all new infections.
Enrollment: 122 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul A. Shuper, PhD, Principal Investigator — Senior Scientist and Section Head
Locations (3):
- Canada (3):
  - Maple Leaf Medical Clinic, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Centre for Addiction and Mental Health, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
Due to the sensitive nature of the data, there is no plan to make IPD available to other researchers. Data will only be accessible to designated research personnel.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Alcohol-focused Brief Intervention | Treatment as Usual
Started | 81 | 41
Completed | 80 | 39
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alcohol-focused Brief Intervention | Treatment as Usual | Total
Number analyzed (Participants) | 81 | 41 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.8 (8.7) | 33.3 (9.3) | 33.6 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 81 | 41 | 122
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 17 | 6 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 51 | 30 | 81
  More than one race | 7 | 1 | 8
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 81 | 41 | 122
AUDIT-C hazardous drinking [Count of Participants; unit: Participants] | 81 | 41 | 122

OUTCOME MEASURES:

1. Primary Outcome: Intervention Feasibility: Intervention Uptake
Description: Intervention uptake will be employed as an indicator of intervention feasibility. Intervention uptake will entail the proportion of eligible, hazardous drinking, PrEP-prescribed MSM who express a willingness to take part in the intervention trial.
Time Frame: At study baseline
Population: 128 were eligible; 122 took part in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Alcohol-focused Brief Intervention
Number analyzed (Participants) | 128
Participants | 122

2. Primary Outcome: Intervention Feasibility: Intervention Completion
Description: Intervention completion will be employed as an indicator of intervention feasibility. This outcome will entail the proportion of participants assigned to the intervention condition who complete the intervention module.
Time Frame: At study baseline
Population: All 81 participants assigned to the intervention condition completed the intervention module.
Measure: Count of Participants; unit: Participants
Arm/Group | Alcohol-focused Brief Intervention
Number analyzed (Participants) | 81
Participants | 81

3. Primary Outcome: Intervention Acceptability
Description: Intervention acceptability will be assessed using a 13-item self-report measure that is comprised of two published scales (references shown below) and three items created by the investigators.
  Bauermeister JA, Pingel ES, Jadwin-Cakmak L, et al. Acceptability and preliminary efficacy of a tailored online HIV/STI testing intervention for young men who have sex with men: the Get Connected! program. AIDS Behav 2015 Oct;19(10):1860-74.
  NDA-NIH. NIMH Data Archive (NDA). 2020. Acceptability of Intervention, Intervention Appropriateness, and Feasibility of Intervention Measure. https://nda.nih.gov/data_structure.html?short_name=aimiamfim01
Time Frame: At 6-months post-baseline
Population: Scales on Items 1-6: 1=Strongly Disagree, 2=Disagree, 3=Somewhat Disagree, 4=Neither Agree or Disagree, 5=Somewhat Agree, 6=Agree, 7=Completely Agree.
  Scales on Items 7-10: 1=Completely Disagree, 2=Disagree, 3=Neither Agree or Disagree, 4=Agree, 5=Completely Agree.
  Scales on Items 11-13: 1=Completely Disagree, 2=Disagree, 3=Neither Agree or Disagree, 4=Agree, 5=Completely Agree.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcohol-focused Brief Intervention
Number analyzed (Participants) | 78
units on a scale
  1. Overall, I was very satisfied with the Personalized Drinking Feedback Report. | 5.72 (1.02)
  2. Using the personalized Drinking Feedback Report was very frustrating. | 2.58 (1.50)
  3. I would recommend the Personalized Drinking Feedback Report to my friends. | 5.27 (1.22)
  4. The Personalized Drinking Feedback Report was easy to use. | 5.76 (0.98)
  5. The Personalized Drinking Feedback Report provided me accurate information. | 5.60 (0.92)
  6. How likely to continue using the Personalized Drinking Feedback Report if it were available? | 4.78 (1.54)
  7. The Personalized Drinking Feedback Report was appealing to me. | 3.47 (0.89)
  8. I liked the Personalized Drinking Feedback Report. | 3.69 (0.74)
  9. I welcomed the Personalized Drinking Feedback Report. | 3.74 (0.81)
  10. The Personalized Drinking Feedback Report met my approval. | 3.85 (0.63)
  11. I benefited from the information provided by the Personalized Drinking Feedback Report. | 3.54 (0.72)
  12. I found the information provided by the Personalized Drinking Feedback Report to be useful. | 3.65 (0.75)
  13. I reduced my drinking as a result of going through the Personalized Drinking Feedback Report. | 2.65 (0.97)

4. Primary Outcome: Alcohol Consumption: Alcohol Use Disorders Identification Test (AUDIT)
Description: Self-report-based Alcohol Use Disorders Identification Test (AUDIT) scores will be compared across baseline, 3-months post-baseline, and 6-months post-baseline sessions. Babor TF, Higgins-Biddle JC, Saunders JB, Monteiro MG, World Health Organization. Dept. of Mental Health and Substance Dependence. The Alcohol Use Disorders Identification Test. Guidelines for Use in Primary Care. 2nd ed. Geneva: World Health Organization; 2001. A cut-off based on AUDIT-C (i.e., AUDIT-consumption) criteria categorizes the presence (i.e., AUDIT-C scores ≥4) or absence (i.e., AUDIT-C scores <4) of hazardous drinking. Minimum and maximum scores of the AUDIT-C are 0 and 12, respectively.
Time Frame: Six months (i.e., baseline, 3-months post-baseline, 6-months post-baseline)
Population: Overall changes in alcohol consumption were evaluated using AUDIT-C hazardous drinking criteria (i.e., AUDIT-C score ≥ 4). Missing values were imputed by controlled multiple imputations.
Measure: Count of Participants; unit: Participants
Arm/Group | Alcohol-focused Brief Intervention | Treatment as Usual
Number analyzed (Participants) | 81 | 41
Participants
  Baseline | 81 | 41
  3-months | 63 | 38
  6-months | 68 | 35

5. Primary Outcome: Alcohol Consumption: Drinks Consumed in a Typical Week
Description: A single self-report question will ask "How many drinks containing alcohol do you have on a typical week when you are drinking?" Responses will be compared across baseline, 3-months post-baseline, and 6-months post-baseline sessions.
Time Frame: Six months (i.e., baseline, 3-months post-baseline, 6-months post-baseline)
Population: Missing values were imputed by controlled multiple imputations.
Measure: Mean (Standard Deviation); unit: Drinks/week
Arm/Group | Alcohol-focused Brief Intervention | Treatment as Usual
Number analyzed (Participants) | 81 | 41
Drinks/week
  Baseline | 8.3 (6.2) | 9.7 (9.0)
  3-months | 8.9 (7.4) | 9.1 (8.0)
  6-months | 9.3 (8.5) | 9.2 (7.9)

6. Primary Outcome: Alcohol Consumption: Maximum Drinks on One Day in the Last 3 Months
Description: A single self-report question will ask "What is the greatest number of drinks you've had on one day in the last 3 months?" Responses will be compared across baseline, 3-months post-baseline, and 6-months post-baseline sessions.
Time Frame: Six months (i.e., baseline, 3-months post-baseline, 6-months post-baseline)
Population: Missing values were imputed by controlled multiple imputations.
Measure: Mean (Standard Deviation); unit: Maximum drinks
Arm/Group | Alcohol-focused Brief Intervention | Treatment as Usual
Number analyzed (Participants) | 81 | 41
Maximum drinks
  Baseline | 7.9 (4.0) | 8.2 (3.7)
  3-months | 7.8 (4.7) | 7.3 (3.4)
  6-months | 7.4 (3.9) | 7.7 (3.2)

7. Primary Outcome: Alcohol Consumption: Phosphatidylethanol (PEth)
Description: PEth levels will be measured from dried blood spot (DBS) samples using liquid chromatography-tandem mass spectrometry to identify hazardous drinking. PEth will be compared across baseline, 3-months post-baseline, and 6-months post-baseline sessions.
Time Frame: Six months (i.e., baseline, 3-months post-baseline, 6-months post-baseline)
Population: PEth levels were dichotomized in accordance with hazardous drinking cut-offs (i.e., PEth ≥ 35 ng/ml). Missing values were imputed by controlled multiple imputations.
Measure: Count of Participants; unit: Participants
Arm/Group | Alcohol-focused Brief Intervention | Treatment as Usual
Number analyzed (Participants) | 81 | 41
Participants
  Baseline | 41 | 23
  3-months | 37 | 18
  6-months | 50 | 27

8. Secondary Outcome: PrEP Adherence: 7-day ACTG-based Measure
Description: Self-reported adherence to PrEP will be assessed using a 7-day, PrEP-focused, ACTG-based adherence measure (the reference for the original, antiretroviral therapy (ART)-focused ACTG measure is shown below). 7-day adherence will be compared across baseline, 3-months post-baseline, and 6-months post-baseline sessions.
  Chesney MA. Ickovics JR. Chambers DB, et al. Self-reported adherence to antiretroviral medications among participants in HIV clinical trials: Tthe AACTG adherence instruments. Patient Care Committee & Adherence Working Group of the Outcomes Committe of the Adult AIDS Clinical Trials Group (AACTG) AIDS Care. 2000;12:255-266.
Time Frame: Six months (i.e., baseline, 3-months post-baseline, 6-months post-baseline)
Population: Missing any PrEP dose during the past 7 days was classified as being non-adherent. Missing values were imputed by controlled multiple imputations.
Measure: Count of Participants; unit: Participants
Arm/Group | Alcohol-focused Brief Intervention | Treatment as Usual
Number analyzed (Participants) | 81 | 41
Participants
  Baseline | 23 | 12
  3-months | 15 | 18
  6-months | 27 | 15

9. Secondary Outcome: PrEP Adherence: Past Month Visual Analog Scale (VAS)
Description: A self-report-based, PrEP-focused visual analog scale (VAS) will be used to assess PrEP adherence over the past month (the reference for the original, antiretroviral therapy (ART)-focused VAS is shown below). Past month adherence will be compared across baseline, 3-months post-baseline, and 6-months post-baseline sessions.
  Amico KR. Fisher WA. Cornman DH, et al. Visual analog scale of ART adherence: Association with 3-day self-report and adherence barriers. J Acquir Immune Defic Syndr. 2006;42:455-459.
Time Frame: Six months (i.e., baseline, 3-months post-baseline, 6-months post-baseline)
Population: Participants who indicated <60% PrEP adherence during the past month were classified as sub-optimally adherent. Missing values were imputed by controlled multiple imputations.
Measure: Count of Participants; unit: Participants
Arm/Group | Alcohol-focused Brief Intervention | Treatment as Usual
Number analyzed (Participants) | 81 | 41
Participants
  Baseline | 6 | 1
  3-months | 2 | 6
  6-months | 6 | 3

10. Secondary Outcome: PrEP Adherence: Tenofovir-diphosphate (TFV-DP) and Emtricitabine-triphosphate Concentrations
Description: Dried blood spots will be assessed for Tenofovir-diphosphate (TFV-DP) and emtricitabine-triphosphate concentrations using validated liquid chromatography tandem mass spectrometry. Concentrations will be compared across baseline, 3-months post-baseline, and 6-months post-baseline sessions.
Time Frame: Six months (i.e., baseline, 3-months post-baseline, 6-months post-baseline)
Population: Tenofovir values were dichotomized to identify any nonadherence (< 1250 fmol/punch). Missing values were imputed by controlled multiple imputations.
Measure: Count of Participants; unit: Participants
Arm/Group | Alcohol-focused Brief Intervention | Treatment as Usual
Number analyzed (Participants) | 81 | 41
Participants
  Baseline | 21 | 15
  3-months | 19 | 14
  6-months | 25 | 18

11. Secondary Outcome: Retention in PrEP Care: PrEP Appointment Attendance
Description: Missed PrEP appointments across the six-month follow-up period will be identified through clinic chart extraction.
Time Frame: Six-month follow-up period
Measure: Count of Participants; unit: Participants
Arm/Group | Alcohol-focused Brief Intervention | Treatment as Usual
Number analyzed (Participants) | 81 | 41
Participants
  Baseline | 6 | 3
  3-months | 1 | 1
  6-months | 2 | 2

12. Secondary Outcome: Condomless Sex
Description: The engagement in condomless anal sex will be assessed using a self-report measure based on an MSM-focused sexual behavior assessment that has been employed in previous trials (see reference below). Condomless sex will be compared across baseline, 3-months post-baseline, and 6-months post-baseline sessions.
  The Explore Team. Effects of a behavioural intervention to reduce acquisition of HIV infection among men who have sex with men: the EXPLORE randomised controlled study. Lancet 2004;364:41-50.
Time Frame: Six months (i.e., baseline, 3-months post-baseline, 6-months post-baseline)
Population: Missing values were imputed by controlled multiple imputations.
Measure: Count of Participants; unit: Participants
Arm/Group | Alcohol-focused Brief Intervention | Treatment as Usual
Number analyzed (Participants) | 81 | 41
Participants
  Baseline | 78 | 38
  3-months | 70 | 37
  6-months | 71 | 33

13. Secondary Outcome: Sexually Transmitted Infection (STI) Incidence
Description: Incident sexually transmitted infections (STIs) during the 6-month follow-up period will be identified through clinic chart extraction.
Time Frame: Six-month follow-up period
Population: Having any STI in the last 3 months was identified through clinic chart extraction.
Measure: Count of Participants; unit: Participants
Arm/Group | Alcohol-focused Brief Intervention | Treatment as Usual
Number analyzed (Participants) | 81 | 41
Participants
  Baseline | 23 | 5
  3-months | 12 | 3
  6-months | 15 | 6

ADVERSE EVENTS:
Time Frame: Data for each participant was collected over 6 month study period.
Arm/Group | Alcohol-focused Brief Intervention | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/41
Other Adverse Events (participants affected / at risk) | 0/81 | 0/41

LIMITATIONS AND CAVEATS:
This was a pilot trial and was therefore not statistically powered to test the effect of the intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-27): https://cdn.clinicaltrials.gov/large-docs/30/NCT05097430/Prot_SAP_000.pdf